CLINICAL TRIAL: NCT05065398
Title: An Open Label， Multicenter Phase II Clinical Trial to Evaluate the Efficacy，Safety and Pharmacokinetics of HLX208 in Advanced Non-small Cell Lung Cancer Patients With BRAF V600 Mutation
Brief Title: A Phase II Clinical Trial to Evaluate HLX208 in Advanced Non-small Cell Lung Cancer Patients With BRAF V600 Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX208-NSCLC201
Record Dates: First submitted 2021-09-09; First posted 2021-10-04 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX208 (Experimental)
  Interventions: Drug: HLX208

INTERVENTIONS:
Drug: HLX208 — 450mg bid, take orally

SUMMARY:
Evaluate the efficacy，safety and pharmacokinetics of HLX208 in advanced non-small cell lung cancer patients with BRAF V600 mutation

ELIGIBILITY:
Inclusion Criteria:

* Age>=18Y
* Good Organ Function
* Expected survival time ≥ 3 months
* advanced BRAF V600 NSCLC that have been diagnosed histologically or cytology and have failed standard treatment or unable to receive, or refusing standard care.
* Previous failure to standard treatment, or insuitability for standard treatment or refuse standard treatment.
* ECOG score 0-2;
* Exclusion Criteria:
* Previous treatment with BRAF inhibitors or MEK inhibitors
* Presence of EGFR mutations or ALK rearrangements (unless disease progression following prior treatment with tyrosine kinase inhibitors).
* Symptomatic brain or meningeal metastases (unless the patient has been on > treatment for 1 months, has no evidence of progress on imaging within 4 weeks prior to initial administration, and tumor-related clinical symptoms are stable).
* Current or former patients with interstitial lung disease;
* Severe active infections requiring systemic anti-infective therapy
* A history of other malignancies within two years, except for cured cervical carcinoma in situ, basal cell carcinoma of the skin, adenocarcinoma in situ of the lung, or tumors that do not require interventional treatment after radical surgery.
* Other anti-tumor treatments, such as chemotherapy, targeted therapy, or radiation therapy (except palliative radiation therapy), may be given during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | from first dose to the last patient was followed up for 6 month
  The number of patients with CR or PR divided by the total number of treated

SECONDARY OUTCOMES:
PFS | the time (month is regarded as the unit) from the first dose to the date of first documented progression or date of death from any cause, whichever came first,through treatment completion, an average of about 1 year
  Progression-free survival
DOR | from the first occurrence of a documented CR or PR (whichever recorded earlier) to the time of first documented disease progression or death (whichever occurs first),through treatment completion, an average of about 1 year
  Duration of response
OS | from the first dose to the time of death due to any cause, an average of about 2 year
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai chest hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol